CLINICAL TRIAL: NCT07209696
Title: Randomized Controlled Evaluation of Storybook and Animation Video as Adjuncts to the Tell-Show-Do Technique in Pediatric Dentistry
Brief Title: Storybook and Animation Video Adjuncts to Tell-Show-Do in Pediatric Dentistry
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Merve Bilmez Selen, PROF LECTURER, Inonu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2024-162
Record Dates: First submitted 2025-09-17; First posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Dental Anxiety; Dental Fear; Child Behavior; Cooperation During Dental Treatment
Keywords: Pediatric Dentistry; Behavior Guidance; Tell-Show-Do; Animation Video Intervention; Jeet Wheel Scale; CFSS-DS; SCAN Index
MeSH Terms: conditions — Child Behavior

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of three parallel groups. The control group will receive the Tell-Show-Do (TSD) technique only. The second group will receive storybook preparation at home followed by TSD. The third group will receive animation video preparation at home followed by TSD. Each participant will remain in the assigned group for the duration of the study.
Who Masked: Outcomes Assessor
Masking Description: The children, parents, and treating dentist were aware of the assigned intervention (storybook, animation video, or Tell-Show-Do only). However, the outcome assessor who rated children's anxiety using the Jeet Wheel scale was blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Tell-Show-Do Only (Control) (Active Comparator): Children in this arm will receive the standard Tell-Show-Do (TSD) behavioral guidance technique before and during dental treatment. No additional preparation such as storybook or animation video will be provided.
  Interventions: Behavioral: Tell-Show-Do
- Storybook + Tell-Show-Do (Experimental): Children in this arm will be prepared at home with a child-friendly storybook that introduces the dental environment, instruments, and treatment steps in an age-appropriate manner. At the clinic, they will then receive the standard Tell-Show-Do (TSD) behavioral guidance technique before and during dental treatment.
  Interventions: Behavioral: Tell-Show-Do; Behavioral: Storybook Preparation
- Animation Video + Tell-Show-Do (Experimental): Children in this arm will be prepared at home with an age-appropriate animation video introducing the dental environment, instruments, and treatment steps. At the clinic, they will then receive the standard Tell-Show-Do (TSD) behavioral guidance technique before and during dental treatment.
  Interventions: Behavioral: Tell-Show-Do; Behavioral: Animation Video Preparation

INTERVENTIONS:
Behavioral: Tell-Show-Do — The conventional behavior guidance technique in pediatric dentistry, where the dentist explains and demonstrates dental procedures before performing them.
Behavioral: Storybook Preparation — Home-based preparation using a child-friendly storybook that introduces the dental visit, instruments, and procedures in simple language and illustrations.
  Arms: Storybook + Tell-Show-Do
Behavioral: Animation Video Preparation — The conventional behavior guidance method where the dentist explains and demonstrates dental procedures before performing them, to reduce anxiety and improve cooperation.
  Arms: Animation Video + Tell-Show-Do

SUMMARY:
This study is designed to evaluate strategies for reducing dental anxiety in pediatric patients. The commonly applied "Tell-Show-Do" method involves explaining and demonstrating dental procedures before they are performed. In this randomized controlled trial, three groups of children will be compared:

Children who receive only the Tell-Show-Do method,

Children who are prepared at home with a storybook prior to receiving the Tell-Show-Do method,

Children who are prepared at home with an animation video prior to receiving the Tell-Show-Do method.

Children's dental anxiety will be assessed using validated behavioral observation scales, including baseline measurement at the first examination, after preparation, and following completion of dental treatment. The study will determine whether the addition of a storybook or an animation video provides greater effectiveness in reducing dental anxiety compared with the Tell-Show-Do method alone.

DETAILED DESCRIPTION:
Dental anxiety is a frequent challenge in pediatric dentistry and can complicate patient cooperation, lead to incomplete treatment, or necessitate the use of general anesthesia. Among the available behavior guidance techniques, the Tell-Show-Do (TSD) method is the most widely applied and has been shown to facilitate children's acceptance of dental procedures. However, recent approaches suggest that additional child-friendly strategies, such as storybooks and animation videos, may further enhance its effectiveness in reducing anxiety and improving cooperation.

This randomized controlled trial aims to evaluate the impact of incorporating a storybook or an animation video in addition to the TSD method on children's dental anxiety and cooperative behavior. Participants will be randomly assigned to one of three groups:

Control group: Tell-Show-Do only.

Storybook group: Children will be prepared at home with a storybook prior to the dental visit, followed by Tell-Show-Do.

Animation video group: Children will be prepared at home with an animation video prior to the dental visit, followed by Tell-Show-Do.

Children's anxiety and cooperation will be assessed at three time points: baseline (first examination), after preparation (before treatment), and after completion of dental treatment. The primary outcome measure will be the Jeet Wheel behavioral observation scale, which provides standardized ratings of children's anxiety and cooperation during dental procedures. In addition, baseline dental fear will be assessed using the Children's Fear Survey Schedule-Dental Subscale (CFSS-DS), and the potential need for general anesthesia will be evaluated with the SCAN Index. These baseline measures will be included as covariates in the statistical analysis to adjust for initial variability in anxiety and treatment requirements.

Data will be analyzed using mixed-effects models to examine the interaction between time (three assessment points) and group (three interventions), while controlling for CFSS-DS and SCAN Index scores. This design will enable comparisons of the relative effectiveness of each intervention independent of baseline differences.

The study is expected to provide new evidence on whether storybook and animation video adjuncts can enhance the effectiveness of the Tell-Show-Do method, offering more child-friendly approaches to reducing dental anxiety in pediatric dental practice.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 4 to 8 years
* Requiring dental treatment in the pediatric dentistry clinic
* Classified as cooperative enough for chairside treatment without mandatory general anesthesia
* Parent or legal guardian able to provide written informed consent
* Child assent obtained where appropriate -

Exclusion Criteria:

* Children with systemic medical conditions that contraindicate routine dental care
* Children with developmental, cognitive, or behavioral disorders that preclude completion of study procedures
* Children requiring urgent dental treatment under general anesthesia or sedation
* Prior exposure to the same storybook or animation video used in the study
* Parents/guardians who decline to provide consent

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in dental anxiety and cooperation measured by the Jeet Wheel Scale | Baseline (Day 1, first examination before intervention) Immediately after preparation, before dental treatment (Day 1, pre-treatment) Immediately after completion of dental treatment (Day 1, post-treatment)
  The Jeet Wheel Scale (JWS) (Chakraborty et al., 2024) is a validated child-friendly tool for evaluating dental anxiety and cooperation. The scale ranges from 1 to 8, represented by expressive emoji faces from Excited (1) to Shouting (8). Lower scores indicate no or minimal anxiety with good cooperation, whereas higher scores indicate severe anxiety and poor cooperation. Children will be asked to select the emoji that best represents their feelings, and the score will be recorded at each time point.

SECONDARY OUTCOMES:
Between-group differences in Jeet Wheel scores after behavioral preparation | Day 1 (Immediately after preparation, before treatment)
  The Jeet Wheel Scale will be assessed immediately after preparation (storybook/video vs. Tell-Show-Do only). Group differences will be analyzed using adjusted statistical models. Scores range from 1 to 8, with higher scores indicating greater anxiety.
Proportion of children with high anxiety at post-treatment (Jeet Wheel score ≥ 4) | Day 1 (Immediately after completion of dental treatment, post-treatment).
  The percentage of participants with a Jeet Wheel score of ≥ 4 will be compared between groups. A higher proportion indicates a greater number of children with clinically relevant anxiety.
Safety and acceptability of behavioral preparations | Throughout the dental visit(s) on Day 1.
  Any adverse events or intolerance related to the behavioral preparation (storybook or video) will be recorded. Examples include refusal to proceed with treatment or discontinuation. Such events are expected to be rare.

OTHER OUTCOMES:
Baseline dental fear assessed by the Children's Fear Survey Schedule-Dental Subscale (CFSS-DS) | Day 1 (Baseline, before intervention).
  The CFSS-DS is a parent-reported measure of children's dental fear. It includes 15 items, each rated 1-5, with total scores ranging from 15 to 75. Higher scores indicate greater dental fear. A score ≥38 indicates clinically significant fear. This score will be collected at baseline and used as a covariate in statistical analysis.
Baseline need for general anesthesia assessed by the SCAN Index | Day 1 (Baseline, before intervention).
  The SCAN Index (Scheduled Care Assessment for Need of General Anesthesia) is used to evaluate the potential need for dental treatment under general anesthesia. Higher scores indicate a greater likelihood of requiring GA. This score will be collected at baseline and included as a covariate in analysis.

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to privacy and confidentiality concerns in pediatric participants.

REFERENCES:
- [Background] Alsaadoon AM, Sulimany AM, Hamdan HM, Murshid EZ. The Use of a Dental Storybook as a Dental Anxiety Reduction Medium among Pediatric Patients: A Randomized Controlled Clinical Trial. Children (Basel). 2022 Mar 1;9(3):328. doi: 10.3390/children9030328. PMID 35327700
- [Background] Barrera-Avalos C, Luraschi R, Acuna-Castillo C, Vidal M, Mella-Torres A, Inostroza-Molina A, Vera R, Vargas S, Hernandez I, Perez C, Vallejos-Vidal E, Valdes D, Imarai M, Reyes-Lopez FE, Sandino AM. Description of Symptoms Caused by the Infection of the SARS-CoV-2 B.1.621 (Mu) Variant in Patients With Complete CoronaVac Vaccination Scheme: First Case Report From Santiago of Chile. Front Public Health. 2022 Mar 21;10:797569. doi: 10.3389/fpubh.2022.797569. eCollection 2022. PMID 35387187
- [Background] Wang Q, Chen S, Li Y, Li P, Wu C, Wu Z, Wu Q, Sun F, Li J, Zheng W, Deng C, Zhang F, Li Y. Positive association of genetic variations in the phospholipase C-like 1 gene with dermatomyositis in Chinese Han. Immunol Res. 2016 Feb;64(1):204-12. doi: 10.1007/s12026-015-8738-x. PMID 26603167
- [Background] Wiley DJ, Grosser S, Qi K, Visscher BR, Beutner K, Strathdee SA, Calhoun B, Palella F, Detels R; Multicenter AIDS Cohort Study Group. Validity of self-reporting of episodes of external genital warts. Clin Infect Dis. 2002 Jul 1;35(1):39-45. doi: 10.1086/340743. Epub 2002 Jun 6. PMID 12060873
- [Background] Thyne SM, Marmor AK, Madden N, Herrick G. Comprehensive asthma management for underserved children. Paediatr Perinat Epidemiol. 2007 Nov;21 Suppl 3:29-34. doi: 10.1111/j.1365-3016.2007.00882.x. PMID 17935573